CLINICAL TRIAL: NCT07252349
Title: Influence of Different Needle Insertion Positions on the Clinical Efficacy of Suture-Fixated Transscleral IOL Implantation Without Knots: A Randomized Controlled Trial
Brief Title: Influence of Different Needle Insertion Positions on the Clinical Efficacy of Suture-Fixated Transscleral IOL Implantation Without Knots
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guangming Jin, Associate Chief Physician, Cataract Department, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025KYPJ136
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Congenital Ectopia Lentis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study adopts a single-blind design, with no blinding of investigators but with blinding of participants and assessors implemented. To reduce bias under the single-blind condition, trial-related personnel involved in participant screening remain blinded, and clinical staff conducting routine ophthalmological examinations as well as data analysts are kept blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group should complete a comprehensive ophthalmic examination at baseline, undergo needle insertion 2.5mm post-limbal during surgery, and receive routine follow-up at 1 week, 1 month, and 3 months postoperatively.
  Interventions: Procedure: Transscleral Suture-Fixated Intraocular Lens Implantation (Suture Needle Insertion at 2.5 mm Posterior to the Limbus)
- compare group (No Intervention): Participants in the intervention group should complete a comprehensive ophthalmic examination at baseline, undergo needle insertion 2mm post-limbal during surgery, and receive routine follow-up at 1 week, 1 month, and 3 months postoperatively.

INTERVENTIONS:
Procedure: Transscleral Suture-Fixated Intraocular Lens Implantation (Suture Needle Insertion at 2.5 mm Posterior to the Limbus) — Participants in the intervention group should complete a comprehensive ophthalmic examination at baseline, undergo needle insertion 2.5mm post-limbal during surgery, and receive routine follow-up at 1 week, 1 month, and 3 months postoperatively.
  Arms: intervention group

SUMMARY:
This is a single-blind, single-center, parallel-group randomized controlled trial with the following objectives: First, researchers aim to compare the clinical efficacy of 2mm and 2.5mm post-limbal needle insertion in sutureless transscleral IOL fixation for patients with congenital ectopia lentis. Second, the goal is to investigate the mean absolute refractive prediction error, IOL tilt and decentration, uncorrected visual acuity (UCVA), best-corrected visual acuity (BCVA), and corneal endothelial cell count at 3 months postoperatively. Third, it intends to explore the incidence of postoperative complications of the two needle insertion positions in this specific surgical method. Finally, this study aims to provide evidence for ophthalmic clinical practice, explore the optimal needle insertion point, and offer more precise and safe surgical plans for patients requiring sutureless transscleral IOL fixation.

DETAILED DESCRIPTION:
This is a professional translation conforming to medical academic writing standards (with unified key terms and specified abbreviation as required):

For patients with insufficient capsular bag support due to congenital developmental abnormalities, trauma, or other reasons, who have indications for intraocular lens (IOL) implantation, IOL suspension surgery is the main surgical method. Sutureless transscleral IOL fixation is one of the commonly used IOL suspension surgeries currently. Compared with traditional transscleral suture fixation, sutureless transscleral IOL fixation can effectively reduce suture-related complications while ensuring safety and effectiveness, with higher surgical safety.

In transscleral IOL fixation, previous studies have commonly used 2mm and 2.5mm post-limbal positions as needle insertion sites. The 2.5mm post-limbal needle insertion point has a smaller mean absolute refractive prediction error and better clinical efficacy postoperatively. As an IOL suspension surgery, differences in needle insertion positions may affect postoperative refractive status, IOL stability, visual outcomes, and other parameters. Although existing literature has evaluated the overall clinical efficacy and safety of sutureless transscleral IOL fixation, to date, no study has systematically compared the clinical efficacy of this commonly used IOL suspension surgery at different needle insertion positions. Therefore, evaluating the impact of different needle insertion positions on surgical outcomes is crucial for optimizing surgical strategies and improving treatment precision.

In this randomized controlled trial, the investigators will systematically investigate the clinical efficacy of 2mm and 2.5mm post-limbal needle insertion points in sutureless transscleral IOL fixation. Through this study, the investigators aim to provide evidence for ophthalmic clinical practice, explore the optimal needle insertion point, and offer more precise and safe surgical plans for patients requiring sutureless transscleral IOL fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 4-18 years (regardless of gender) who meet the indications for transscleral suture-fixated intraocular lens implantation
2. Patients who can complete a follow-up period of at least 3 months after surgery;
3. Patients or their legal guardians who provide informed consent to participate in this study.

Exclusion Criteria:

1. Patients with concurent secondary qlaucoma, retinal detachment, strabismus, or other relevant ocular complications (excludingrefractive errors);
2. Patients participating in other trials that may affect the results of this study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Refractive Predictive Error of Patients at the 3-month Postoperative Follow-up | 3-month Postoperative Follow-up
  Case report form records

SECONDARY OUTCOMES:
Uncorrected Visual Acuity (UCVA) and Best-Corrected Visual Acuity (BCVA) of Patients at the 3-Month Postoperative Follow-up | 3-month Postoperative Follow-up
  Measured using the EDTRS chart
lOL Tilt and Decentration in Patients at the 3-Month Postoperative Follow-up | 3-month Postoperative Follow-up
  Measured by the Casia 2 AS-OCT Instrument
Corneal Endothelial Cell Count of Patients at the 3-Month Postoperative Follow-up | 3-month Postoperative Follow-up
  Measured using a corneal endothelial microscope
Incidence of Postoperative Complications at the 3-Month Postoperative Follow-up | 3-month Postoperative Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Danying Zheng, Study Chair — Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, ZhongshanOphthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual SodGuangzhou, Guangdong; Guangming Jin, Principal Investigator — Guangdong Provincial Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology, ZhongshanOphthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology and Visual ScienceGuangzhou, Guangdong
Locations (1):
- Clinical Research Center for Ocular Diseases, State Key Laboratory of Ophthalmology,Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangdong Provincial Key Laboratory of Ophthalmology andVisual Science, Guangzhou, Guangdong, Guangdong, Province, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code

REFERENCES:
- [Result] Qu Y, Duan P, Huo S, Li F, Li J. Sutured Intrascleral Posterior Chamber Intraocular Lens Fixation with Ciliary Sulcus Location Guided by Ultrasonic Biological Microscopy: A Retrospective Analysis of Anatomical and Refractive Outcome. J Ophthalmol. 2020 Jun 4;2020:5843410. doi: 10.1155/2020/5843410. eCollection 2020. PMID 32587761
- [Result] Kim J, Lee PY, Park MS, Cho BJ, Kwon S. Comparison of outcomes between modified double-flanged sutureless scleral fixation and conventional sutured scleral fixation. Sci Rep. 2024 Jul 12;14(1):16111. doi: 10.1038/s41598-024-66762-y. PMID 38997328
- [Result] Yoon EG, Eom Y, Woo M, Jeon HS, Kim SJ, Song JS, Kim HM. Clinical Outcomes of Intrascleral Fixation of Intraocular Lens Compared to Ciliary Sulcus Implantation and Transscleral Fixation. Korean J Ophthalmol. 2023 Apr;37(2):128-136. doi: 10.3341/kjo.2022.0093. Epub 2023 Feb 9. PMID 36758538
- [Result] Dubinsky-Pertzov B, Mahler OS, Hecht I, Shemer A, Or L, Gazit I, Pras E, Einan-Lifshitz A. Accuracy of Intraocular Lens Calculation Formulas for the Four-Flanged Fixation Technique in Eyes With No Capsular Support. J Refract Surg. 2022 Oct;38(10):668-673. doi: 10.3928/1081597X-20220919-01. Epub 2022 Oct 1. PMID 36214349
- [Result] Leuzinger-Dias M, Lima-Fontes M, Rodrigues R, Oliveira-Ferreira C, Madeira C, Falcao-Reis F, Fernandes V, Rocha-Sousa A, Falcao M. Scleral Fixation of Akreos AO60 Intraocular Lens Using Gore-Tex Suture: An Eye on Visual Outcomes and Postoperative Complications. J Ophthalmol. 2021 Dec 20;2021:9349323. doi: 10.1155/2021/9349323. eCollection 2021. PMID 34966559
- [Result] Micheletti JM, Weber N, McCauley MB, Doe EA, Coffee RE, Caplan MB. Punch and rescue technique for scleral fixation of dislocated single-piece intraocular lenses. J Cataract Refract Surg. 2022 Feb 1;48(2):247-250. doi: 10.1097/j.jcrs.0000000000000845. PMID 34670946
- [Result] Zeilinger J, Kronschlager M, Schlatter A, Ruiss M, Bayer N, Findl O. Influence of Sutureless Scleral Fixation Techniques With 3-Piece Intraocular Lenses on Dislocation Force. Am J Ophthalmol. 2024 Aug;264:229-234. doi: 10.1016/j.ajo.2024.03.001. Epub 2024 Mar 10. PMID 38461946
- [Result] Shi J, Zong Y, Wu K, Jiang C. Simplified Technique for Correcting Intraocular Lens Decentration in Scleral-Sutured Fixation Surgery. Retina. 2025 Jan 17. doi: 10.1097/IAE.0000000000004401. Online ahead of print. PMID 39841916
- [Result] Lee KRCK, Fung AT. Four-point subconjunctival scleral fixation technique using Gore-Tex suture. Clin Exp Ophthalmol. 2021 May;49(4):397-399. doi: 10.1111/ceo.13938. Epub 2021 May 11. No abstract available. PMID 33913234
- [Result] Dogan L, Edhem Yilmaz I. Quaternary Knot Technique: Suture Knot Burial without Scleral Flap or Incision for Trans-scleral Fixation. J Ophthalmic Vis Res. 2023 Jul 28;18(3):342-347. doi: 10.18502/jovr.v18i3.13784. eCollection 2023 Jul-Sep. PMID 37600913
- [Result] Czajka MP, Frajdenberg A, Johansson B. Technique for Sutured Scleral Fixation of One-Piece Hydrophobic Acrylic Intraocular Lenses Dislocated Into the Vitreous. Retina. 2023 Aug 1;43(8):1413-1416. doi: 10.1097/IAE.0000000000003008. PMID 33149099
- [Result] Byun Z, Kim DI, Kong M. LONG-TERM ANALYSIS OF INTRASCLERAL FIXATION OF INTRAOCULAR LENS: Trocar-Cannula-Based Sutureless Intrascleral Fixation Versus Sutured Scleral Fixation. Retina. 2023 May 1;43(5):815-822. doi: 10.1097/IAE.0000000000003721. PMID 36728892
- [Result] Choi HJ, Kwon OW, Byeon SH, Song JH. Clinical outcomes of combined pars plana vitrectomy and scleral fixation of the intraocular lens with a suspension bridge method in eyes with aphakia or insufficient capsular support. Acta Ophthalmol. 2021 Nov;99(7):e1006-e1012. doi: 10.1111/aos.14758. Epub 2021 Jan 9. PMID 33421312